CLINICAL TRIAL: NCT02935868
Title: Periodontal and Salivary Evaluation of a Sample of Type 1 Diabetes Mellitus Patients in Brazil
Brief Title: Periodontal and Salivary Evaluation of Type 1 Diabetes Mellitus Patients
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carla Andreotti Damante, Associate professor, University of Sao Paulo
Other Study IDs: Bauru School of Dentistry
Record Dates: First submitted 2016-09-29; First posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 1; Periodontal Diseases
Keywords: Saliva
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Test group: Patients with Type 1 diabetes mellitus
- Control Group: Patients without systemic diseases

SUMMARY:
Diabetes Mellitus is a risk factor for periodontal disease increasing its prevalence, extension and severity. Periodontal disease is considered the sixth complication of diabetes. There is a global epidemic of diabetes, including an increase of incidence of type 1 diabetes in younger patients. Thus, the aim of this observational study was to evaluate the periodontal and salivary condition of a sample of patients with type 1 diabetes of a brazillian city.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose of Type 1 diabetes mellitus
* Age between 18 and 35 years old
* Presenting on tooth per quadrant

Exclusion Criteria:

* Diagnose of Type 2 diabetes mellitus
* Edentulous patients
* Other systemic diseases

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Test Group: Patients diagnosed with Type 1 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Periodontal disease (gingivitis and periodontitis) measured by a periodontal probe and classified according to severity | one day
  Severe periodontitis was defined by the presence of ≥ 2 interproximal sites in different teeth with CAL (clinical attachment level) ≥ 6mm and ≥1 interproximal site with PPD (periodontal probing depth) ≥5mm. Moderate periodontitis was defined by the presence of ≥ 2 interproximal sites in different teeth with CAL ≥ 4mm or ≥ 2 interproximal sites in different teeth with PPD ≥5mm. Mild periodontitis was defined as ≥ 2 interproximal sites in different teeth with ≥ 3 mm CAL and ≥ 2 interproximal sites in different teeth with ≥ 4 mm PPD or at least 1 site with PPD ≥ 5 mm (20,21). Gingivitis was determined as follows: Subjects were considered healthy if presented PPD ≤3mm/BOP (bleeding on probing) extent scores < 10% and with gingivitis if presented PPD ≤3mm/ BOP extent scores >10%.
Salivary pH and buffering Capacity - collection of stimulated saliva in 10 minutes and measurement of acidity with a pHmeter | one day
  Normal Salivary pH = 6 to 7. Buffering capacity: ≥ 5.6 were considered as ''high'', ranging from 4.1 to 5.5 were labelled as ''medium'' and those ≤4 were defined as ''low''
Salivary glucose - collection of stimulated saliva in 10 minutes and measurement with a colorimetric kit | one day
  Salivary glucose is measured by a colorimetric kit and the values are converted and presented as mg/dL. There are no reference value for this measurement. The analysis is done by means of correlation to blood glucose levels in mg/dL.
Salivary peroxidase - collection of stimulated saliva in 10 minutes, measurement by a spectrophotometer. | one day
  The activity of salivary peroxidase is presented in Units/mg. The detection of activity of these enzymes is associated to periodontal disease.

SECONDARY OUTCOMES:
Plaque index - measured by visual observation and classification in scores (1 for presence, 0 for absence) | One day
  Plaque index (PI) will be registered as scores (1 for presence, 0 for absence). For control group a plaque index of 15% is considered normal.

CONTACTS AND LOCATIONS:
Locations (1):
- Bauru School of Dentistry, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aren G, Sepet E, Ozdemir D, Dinccag N, Guvener B, Firatli E. Periodontal health, salivary status, and metabolic control in children with type 1 diabetes mellitus. J Periodontol. 2003 Dec;74(12):1789-95. doi: 10.1902/jop.2003.74.12.1789. PMID 14974821
- See also: Master Thesis in Portuguese - abstract in english — http://www.teses.usp.br/teses/disponiveis/25/25146/tde-26042016-102416/pt-br.php